CLINICAL TRIAL: NCT03812380
Title: Averting Complications of Proton Pump Inhibitor Therapy by Effervescent Calcium Magnesium Citrate
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to a severe decrease in enrollment over the years 2020 and 2021. The major obstacle which hindered participation of subjects was the COVID-19 pandemic. Research was halted. Remaining study patients were withdrawn.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Khashayar Sakhaee, Chief, Division of Mineral Metabolism; Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU 042018-078
Record Dates: First submitted 2018-05-24; First posted 2019-01-23 (Actual); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Osteoporosis; Hypomagnesemia
Keywords: Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — effervescent calcium magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To provide adequate blinding, each medication sachet will be labelled with the study name, IRB number, principal investigator's name, expiration date and identification number of the study subject. Labels will be applied to the appropriate medication sachets once the subject has been randomized and assigned to a treatment group. Labelling of the sachets will be done by personnel who are not engaged in patient care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EffCaMgCit (Experimental): 19 meq or 380 mg calcium, 10 meq (122 mg) magnesium, and 50 meq total citrate; designed to be added to 6 oz water for 1-2 minutes, to be dissolved/suspended before swallowing. Each sachet of EffCaMgCit will contain 400 units of vitamin D.
  Interventions: Drug: EffCaMgCit
- Placebo (Placebo Comparator): Each sachet of Placebo will contain microcrystalline cellulose, but no calcium, magnesium or citrate. Placebo will be added to 6 oz water for 1-2 minutes, to be dissolved/suspended before swallowing. The placebo will contain 400 units of vitamin D.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EffCaMgCit — Each sachet of EffCaMgCit will contain 19 meq or 380 mg calcium, 10 meq (122 mg) magnesium, and 50 meq total citrate.
  Other Names: Effervescent calcium magnesium citrate
  Arms: EffCaMgCit
Other: Placebo — Each sachet of Placebo will contain microcrystalline cellulose, but no calcium, magnesium or citrate. Placebo will be added to 6 oz water for 1-2 minutes, to be dissolved/suspended before swallowing. The placebo will contain 400 units of vitamin D.
  Arms: Placebo

SUMMARY:
Proton pump inhibitors (PPIs) are widely used for the control of gastric ulcer-gastritis, erosive esophagitis (gastroesophageal reflux disease), peptic ulcer disease (duodenal ulcer), and heartburn. Despite their efficacy, their use has been implicated in possibly causing fragility fractures (osteoporosis), hypomagnesemia (magnesium deficiency) and increased risk of chronic kidney disease (CKD). The current trial represents the investigators' ongoing effort to discern whether these complications could be averted by effervescent calcium magnesium citrate (EffCaMgCit).

DETAILED DESCRIPTION:
In a single-dose bioavailability study, the investigators showed previously that provision of calcium and magnesium in a soluble form as EffCaMgCit improved intestinal absorption of calcium and magnesium and suppressed parathyroid function during PPI treatment, compared with calcium carbonate. In a multidosing trial with esomeprazole 40 mg/day for 28 days, EffCaMgCit suppressed parathyroid function and bone turnover, and increased serum and urinary magnesium, compared with placebo. Moreover, EffCaMgCit co-administered with PPI conferred an alkali load, and averted apparent acid load conferred by PPI (when given with placebo).

In the current proposal, the investigators wish to conduct a 2-year treatment trial, directed at obtaining more definitive evidence that EffCaMgCit overcomes all three complications of PPI.

Aim 1. To test the hypothesis that EffCaMgCit would prevent/treat osteoporosis, by suppressing parathyroid function and bone resorption, thereby stabilizing bone mineral density (BMD). The critical endpoint will be BMD. Secondary endpoints will be serum PTH and C-terminal telopeptide (CTX).

Aim 2. To test the hypothesis that EffCaMgCit would prevent/treat hypomagnesemia/magnesium deficiency, by providing bioavailable magnesium. The critical endpoint will be fractional excretion of magnesium (FEMg) and free muscle magnesium by MRS. Secondary endpoints will be serum and urinary magnesium.

Aim 3. To test the hypothesis that EffCaMgCit would reduce the risk of CKD during PPI use by averting putative hypomagnesemia/magnesium deficiency and neutralizing acid load. The investigators propose that PPI causes hypomagnesemia/magnesium deficiency and confers an acid load, - factors implicated for incident CKD and its progression. EffCaMgCit is expected to avert incident CKD by providing bioavailable magnesium and alkali load. Critical endpoints will be endogenous creatinine clearance, FEMg, free muscle magnesium and acid-base status.

ELIGIBILITY:
Inclusion Criteria:

* Must have taken PPI (omeprazole or equivalent ≥ 20 mg/day, ≥ three times per week, for at least 2 months)
* Expected to continue at a similar dosage
* Stage 1 hypertension (with systolic blood pressure <140 and diastolic <90)
* controlled diabetes mellitus Type II with HbA1C less than 7%

Exclusion Criteria:

* end-stage renal failure on dialysis
* hypercalcemia
* hypophosphatemia (serum P < 2.5 mg/dL)
* hypertension stage 2 or higher
* diabetes Type II with HbA1C ≥ 7%
* treatment with adrenocorticosteroids, diuretics, non-steroidal anti-inflammatory agents
* regular dose of magnesium supplements, bisphosphonate, teriparatide, denosumab or selective estrogen receptor modulators.

Inclusion/exclusion of other drugs or conditions will be considered on an individual basis.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Sakhaee, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 62 participants enrolled, only 44 met the inclusion criteria and were randomized to the treatment.
Period: Overall Study
Arm/Group | EffCaMgCit | Placebo
Started | 22 | 22
Completed | 0 | 1
Not Completed | 22 | 21
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Early termination of study | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EffCaMgCit | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 16 | 28
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) T-Score at 2 Years
Description: Change from baseline in bone mineral density (BMD) T-Score at 2 years as measured by dual photon absorptiometry. The range, as defined by the World Health Organization (WHO), for T-Score is: -1 and above = Normal, Between -1 and -2.5 = Osteopenia, -2.5 and below = osteoporosis.
Time Frame: Baseline and 2 years
Population: Because of severe enrollment difficulty due to COVID-19 restrictions and consequently a suspension of research activities, this study was terminated early. Only one subject completed the full two year duration for which data are summarized here.
Measure: Number; unit: T-Score
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
T-Score
  L2-L4 T-Score |  | -0.4
  Femoral Neck T-Score |  | -1.0
  Total Hip T-Score |  | -0.7
  Radial 1/3rd T-Score |  | -0.3

2. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) Z-Score at 2 Years
Description: Change from baseline in bone mineral density (BMD) Z-score at 2 years as measured by dual photon absorptiometry. Outcome is considered positive if the Z Score after two years of treatment becomes less negative (less than -2). There is no specific score range for the Z Score.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: Z-Score
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
Z-Score
  L2L4 Z-Score |  | -0.1
  Femoral Neck Z-Score |  | -0.8
  Total Hip Z-Score |  | -0.7
  Radial 1/3rd Z-Score |  | -0.1

3. Primary Outcome: Change From Baseline in the Fractional Excretion of Magnesium (FEMg) at 2 Years
Description: Change from baseline in the fractional excretion of magnesium (FEMg) at 2 years as measured by the ratio of magnesium clearance and creatinine clearance, using 24-h urinary magnesium and creatinine and corresponding serum magnesium and creatinine obtained post meal/load.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: percentage
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
percentage |  | -1.0

4. Primary Outcome: Change From Baseline in Free Muscle Magnesium at 2 Years
Description: Change From baseline in free muscle magnesium at 2 years as assessed by measuring intracellular Mg in a calf muscle, by using 31P (Phosphorous) magnetic resonance spectroscopy (MRS).
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: mmol/L
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
mmol/L |  | -0.044

5. Primary Outcome: Change From Baseline in Endogenous Creatinine Clearance at 2 Years
Description: Change from baseline in endogenous creatinine clearance at 2 years will be measured. Endogenous creatinine clearance will be obtained by using 24-h urinary creatinine and post-meal/load venous blood sample ((uCr, mg/24hr) / (sCr,mg/dL * 14.4))
Time Frame: Baseline and 2 years
Population: Because of severe decrease in enrolled participants due to COVID-19 restrictions and consequently a suspension of research activities resulted in the early termination of this study. Only 1 subject completed the 2 year timepoint for which the data is summarized here.
Measure: Number; unit: ml/min
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
ml/min |  | 13

6. Secondary Outcome: Change From Baseline in Serum Parathyroid Function (PTH) at 2 Years
Description: Change from baseline in serum parathyroid function (PTH) at 2 years will be measured by Biomerica Intact-PTH ELISA.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: pg/ml
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
pg/ml |  | 75

7. Secondary Outcome: Change From Baseline in Serum Bone Resorption Marker C-terminal Telopeptide (CTX) at 2 Years
Description: Change from baseline in serum bone resorption marker C-terminal telopeptide (CTX) at 2 years will be measured by lab finding utilizing ELISA CTX-I (CrossLaps).
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: ng/ml
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
ng/ml |  | 0.15

8. Secondary Outcome: Change From Baseline in Serum Magnesium at 2 Years
Description: Change from baseline in serum magnesium at 2 years will be measured by ion selective electrode.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: mg/dL
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
mg/dL |  | 0.2

9. Secondary Outcome: Change From Baseline in Urine Magnesium at 2 Years
Description: Change from baseline in urine magnesium at 2 years was measured by by atomic absorption.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: mg/day
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
mg/day |  | -8

10. Secondary Outcome: Change From Baseline in Serum Bicarbonate at 2 Years
Description: Change from baseline in serum bicarbonate at 2 years will be measured to see improvement in acid based status in lowering kidney function impairment.
Time Frame: Baseline and 2 years
Population: as for outcome 1
Measure: Number; unit: mmol/L
Arm/Group | EffCaMgCit | Placebo
Number analyzed (Participants) | 0 | 1
mmol/L |  | -2

ADVERSE EVENTS:
Time Frame: From the participant's first dose at baseline (0 month) to the end of 24 months
Description: A severe decrease in the enrolled participants due to COVID restrictions and consequently a suspension of research activities resulted in the early termination of this study.
Arm/Group | EffCaMgCit | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EffCaMgCit (N=22) | Placebo (N=22)
Gas, smelly gas and bloating (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03812380/Prot_SAP_000.pdf